CLINICAL TRIAL: NCT02370147
Title: The Effect of Very Brief Smoking Reduction Intervention in Smokers Who Having no Intention to Quit: Study Protocol for a Randomized Controlled Trial
Brief Title: Very Brief Smoking Reduction Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yao He, Institute of Geriatrics, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ChinaPLAGHW
Record Dates: First submitted 2015-02-10; First posted 2015-02-24 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Smoking Cessation
Keywords: smoking reduction intervention; no intention to quit; randomized controlled trial; telephone follow-up intervention
MeSH Terms: conditions — Smoking Cessation | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smoking reduction intervention arm (Experimental): Smoking reduction intervention arm (SRI) consisting of a minimal face-to-face individual smoking reduction intervention lasted for about one minute, and five follow-up interventions lasted for about one minute each.
  Interventions: Behavioral: Smoking reduction intervention
- Control arm (Active Comparator): Control arm (UC) consisting of a brief face-to-face individual exercise and dietetic advices lasted for the same intervention time as SRI, and five follow-up interventions lasted for about one minute each with different intervention contents.
  Interventions: Behavioral: Exercise and diet advice control

INTERVENTIONS:
Behavioral: Smoking reduction intervention — Smokers was informed that many harmful effects were proved to be related with smoking, such as cancer, coronary heart disease, respiratory disease and many other health problems, and one out of two smokers will be killed by smoking. Smokers will be advised to reduce smoking consumption for at least half of their total consumption in the next month. Finally, all smokers were warned to keep in mind that the current attempt to reduce smoking is an intermediate step before the complete cessation.
  Arms: Smoking reduction intervention arm
Behavioral: Exercise and diet advice control — Smokers will be asked to do regular activities for three or four times per week, and to have a healthy and balanced diet, having more fruit and vegetables which are rich in vitamins, high in nutrition yet low in calories. In the whole process, advises will not refer to smoking cessation or smoking reduction.
  Arms: Control arm

SUMMARY:
A two-arm randomized controlled trial for smokers who are not intent to quit smoking will be proposed in outpatient department clinics of People's Liberation Army General Hospital in Beijing, China. Smoking reduction intervention arm (SRI) consisting of a very brief face-to-face individual smoking reduction intervention lasted about one minute, and five follow-up interventions lasted for about minute each. Control arm (EDA) consisting of a very brief face-to-face individual exercise and dietetic advices lasted for the same intervention time as SRI, and also five follow-up interventions lasted for one minute each with different intervention contents.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years old;
2. Smoked more than 10 cigarettes per day in the past month.
3. Have no intent to smoking cessation now.
4. Agreed to participate in the follow-up, offer telephone number and signed an informed consent form.

Exclusion Criteria:

1. Smoked less than 10 cigarettes per day in the past month.
2. Had some diseases that let the physician think that it would be unethical not to advise him to quit smoking as soon as possible.
3. Cognitively impaired (such as those with deafness or who could not understand and complete the questionnaire reliably).
4. Pregnant females.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
self-reported 7-day point prevalence quit rate | at 12 months follow-up
prolonged abstinence quit rate | at 12 months follow-up

SECONDARY OUTCOMES:
smoking reduction rates | baseline and at 12 months follow-up
  number of cigarettes smoked per day reduced at least 50%

REFERENCES:
- [Derived] Wu L, He Y, Jiang B, Zhang D, Tian H, Zuo F, Lam TH, Cheung YT. The effect of a very brief smoking-reduction intervention in smokers who have no intention to quit: study protocol for a randomized controlled trial. BMC Public Health. 2015 Apr 25;15:418. doi: 10.1186/s12889-015-1749-7. PMID 25944023